CLINICAL TRIAL: NCT00332280
Title: A Prospective, Randomised, Multicenter Phase II/III Clinical Trial to Evaluate the Clinical Benefit Response in Cancer Patients With Advanced Disease With AMT Versus Placebo
Brief Title: Study to Evaluate the Clinical Benefit Response in Cancer Patients With Advanced Disease With AMT2003 Versus Placebo
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy. Stopped at first interim evaluation point
Sponsor: Auron Healthcare GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMT/P2CA/001; LC003AURON2005
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Gastrointestinal Cancer; Prostate Cancer; Genital Neoplasms, Female
Keywords: solid tumors; clinical benefit; quality of life; esophageal cancer; colon cancer; pancreatic cancer; gastric cancer; liver cancer; gall bladder cancer; prostate cancer; gynecological cancer; lung cancer; Tumors of GI tract, prostate and gynaecological
MeSH Terms: conditions — Gastrointestinal Neoplasms; Prostatic Neoplasms; Genital Neoplasms, Female; Esophageal Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Liver Neoplasms; Gallbladder Neoplasms; Lung Neoplasms

ARMS (1):
- AMT2003 (Experimental)
  Interventions: Drug: AMT2003

INTERVENTIONS:
Drug: AMT2003

SUMMARY:
The purpose of the study is to evaluate the efficacy and the safety of AMT2003 in cancer patients with advanced disease.

The primary evaluation criterion is clinical benefit response.

DETAILED DESCRIPTION:
The study will include patients with a variety of solid tumors (i.e. esophageal, colon, pancreatic, bronchial, gastric, hepatocellular, gall bladder, prostate and gynaecological carcinomas.)

The clinical benefit response - CBR, is an end point that provides a clinical measure for symptom improvement in patients. The key evaluation parameters for CBR will be assessment of pain, the ability to perform daily activities and weight change.

ELIGIBILITY:
Inclusion Criteria:

* Cancer confirmed by histology or cytology
* At least one measurable lesion
* Advanced disease refractory to standard therapy or for which no standard therapy exists
* Life expectancy at least 3 months

Exclusion Criteria:

* Known secondary neoplasia or central nervous system (CNS) metastases, acute or chronic leukemia, lymphoma or multiple myeloma
* Body weight below 45 kg
* Female patients who are pregnant or breast feeding or adults of reproductive potential not employing effective birth control methods
* Concurrent severe or uncontrolled medical disease
* Acute or chronic liver disease
* Confirmed diagnosis of HIV
* Insulin dependent diabetes mellitus/abnormal glucose tolerance test (GTT)/latent diabetes mellitus type I or II
* Chemotherapy or radiotherapy less than 4 weeks prior to entry
* Surgery less than 2 weeks prior to entry (or not recovered from effects of surgery)
* Participation in a clinical trial less than 30 days prior to entry into this study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-05; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Improvement in clinical benefit response | Jan 2010

SECONDARY OUTCOMES:
Progression free survival | Jan 2010
Overall survival | Jan 2010
Overall response rate | 2010
Duration of response | January 2010
Quality of life (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire [EORTC QLQ-C30]) | Jan 2010
Safety and tolerability | Jan 2010

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Drevs, PD Dr. Med, Principal Investigator — Clinic SanaFontis
Locations (2):
- Klinicki Centar Univerziteta Sarajevo - Klinika za gastroenterohepatologiju, Sarajevo, Bosnia and Herzegovina
- Clinic SanaFontis, Freiburg im Breisgau, Germany

REFERENCES:
- See also: Alpinia Institute now legally responsible for the study — http://www.alpiniainstitute.com